CLINICAL TRIAL: NCT06606704
Title: Effects of Resistance-band Training and Creatine Supplementation in Healthy Older Adults
Brief Title: Effects of Resistance-band Training and Creatine Supplementation Strategies in Healthy Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Iovate Health Sciences International Inc (Industry)
Responsible Party: Principal Investigator, Darren Candow, Professor, University of Regina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 853
Record Dates: First submitted 2024-09-16; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Aging
Keywords: Aging; Creatine; Resistance-Bands; Muscle; Strength

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Creatine Bolus 5 (Experimental)
  Interventions: Dietary Supplement: Creatine Bolus 5
- Creatine Bolus 3 (Experimental)
  Interventions: Dietary Supplement: Creatine Bolus 3
- Creatine Intermittent 5 (Experimental)
  Interventions: Dietary Supplement: Creatine Intermittent 5
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine Bolus 5 — (Serving 1: 5 grams of creatine + 3 grams of placebo in the morning; Serving 2: 8 grams of placebo at least 6 hours after Serving 1).
  Arms: Creatine Bolus 5
Dietary Supplement: Creatine Bolus 3 — (Serving 1: 3 grams of creatine + 5 grams of placebo in the morning; Serving 2: 8 grams of placebo at least 6 hours after Serving 1).
  Arms: Creatine Bolus 3
Dietary Supplement: Creatine Intermittent 5 — (Serving 1: 2.5 grams of creatine + 5.5 grams of placebo in the morning, Serving 2: 2.5 grams of creatine + 5.5 grams of placebo at least 6 hours after Serving 1).
  Arms: Creatine Intermittent 5
Dietary Supplement: Placebo — (Serving: 8 grams of placebo in the morning; Servings 2: 8 grams of placebo at least 6 hours after Serving 1).
  Arms: Placebo

SUMMARY:
The primary purpose is to compare the effects of creatine supplementation (bolus ingestion of 5 grams vs. 3 grams) during 16 weeks of resistance-band training on measures of body composition (i.e., whole-body lean tissue mass, total body water), arm and leg muscle thickness (growth), muscle performance (i.e., power, strength, endurance) and functional ability (i.e., walking speed, balance).

A secondary purpose of this research is to examine the effects of bolus ingestion of creatine (5 grams) compared to intermittent ingestion of creatine (2 x 2.5 grams) during 16 weeks of resistance-band training on measures of body composition (i.e., whole-body lean tissue mass, total body water), arm and leg muscle thickness (growth), muscle performance (i.e., power, strength, endurance) and functional ability (i.e., walking speed, balance).

DETAILED DESCRIPTION:
Resistance-band training is safe, conveient, easy-to-use, eliminates potential barriers to exercise participation (i.e., lack of transportation to and from commercial training facilities) and results in high exercise compliance and adherence. Further, resistance-band training results in similar improvements in muscle performance and functional ability compared to traditional resistance-type training using free-weights and machines.

Creatine is a naturally occurring nitrogen-containing compound produced in the body in the liver and brain and can also be found in food products such as red meat and seafood or through commercially available manufactured creatine products.

Evidence-based research shows that creatine supplementation, when ingested during a resistance exercise training program, improves measures of lean mass and muscle growth, muscle performance and functional ability. However, the optimal creatine supplementation protocol to achieve these benefits is unknown.

ELIGIBILITY:
Inclusion Criteria:

* if you are 50 years of age and older
* if you have not been performing more than 1 resistance training session per week for the past 6 weeks or more.

Exclusion Criteria:

* if you have taken creatine supplements within 30 days prior to the start of the study
* if you have pre-existing allergies to the placebo (corn-starch maltodextrin).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Whole-body lean mass (kg) | baseline, week 16
  Bioelectrical impedance analysis
Muscle Hypertrophy (cm) | baseline, week 16
  B-mode ultrasound
Strength (kg) | baseline, week 16
  1-repetition maximum leg press and chest press
Endurance (number of repetitions to fatigue) | baseline, week 16
  Leg press and chest press
Power (feet) | baseline, week 16
  medicine ball throw
Balance (Centre of Pressure) | baseline, week 16
  Force Plate
Gait Speed (meters) | baseline, week 16
  Walking distance

CONTACTS AND LOCATIONS:
Overall Officials: Darren Candow, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No